CLINICAL TRIAL: NCT00373100
Title: The Efficacy of Zinc as Adjunct Therapy in the Treatment of Severe Pneumonia in Children Admitted to Mulago Hospital, Uganda.
Brief Title: The Efficacy of Zinc as Adjunct Therapy in the Treatment of Severe Pneumonia in Children
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Makerere University (Other)
Responsible Party: James K Tumwine, Department of Paediatrics and Child Health Makerere University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HD1120041349X
Record Dates: First submitted 2006-09-06; First posted 2006-09-07 (Estimated); Last update posted 2009-07-07 (Estimated); Status verified 2009-07

CONDITIONS: Pneumonia
Keywords: Zinc; placebo; severe pneumonia; children
MeSH Terms: conditions — Pneumonia | interventions — Zinc Acetate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Zinc (Experimental): Zinc acetate
  Interventions: Drug: Zinc acetate
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Zinc acetate
  Arms: Zinc
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
Pneumonia is a leading cause of morbidity and mortality in children in developing countries. Zinc deficiency leads to impairment in tissue repair and immunodeficiency in children.At least two randomised controlled trials have shown that zinc supplementation improves the outcome of severe pneumonia in children (reducing duration of hospital stay and complications related to pneumonia).

However, there are conflicting results from other randomised controlled trials about its efficacy in children with pneumonia.The purpose of the current study is to determine the efficacy of zinc as adjunct therapy for in severe pneumonia in children aged 6-59 months. We hypothesize that the proportion of children who recover from severe pneumonia following zinc adjunct therapy [(10 mg once daily for seven days) for children aged <12 months and 20 mg daily for children aged ≥12 months]will be higher than the proportion of children who recover from placebo therapy.

DETAILED DESCRIPTION:
Zinc deficiency is a global nutritional problem affecting people with a low socioeconomic status in developing and developed countries. There is a high prevalence of zinc deficiency in Uganda as documented by Bitarakwate et al.Two clinical studies have shown that zinc supplementation improves the outcome of severe pneumonia in children by reducing duration of hospital stay and complications related to pneumonia. However, there are conflicting results from some previous studies about its usefulness in patients with pneumonia.

The objective of this study is to determine the effect of zinc supplement as adjunct therapy in the treatment of severe pneumonia in children less than five years admitted to Mulago hospital, Kampala, Uganda.

This will be a randomized, double-blinded, placebo-controlled trial of zinc adjucnt therapy. Three hundred and twenty eight children with severe pneumonia will be randomised to receive either zinc (a daily dose of 20 mg for children more than one of age and 10mg for those less than one year or placebo once daily for seven days.

The primary outcome will be Time taken to :normalisation of respiratory rate, temperature and oxygen saturation.

Secondary outcome:Proportion of study children who will die during the follow up period,Proportion of children who develop drug adverse effects data will be analysed using Kaplan Meir survival curves.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 6- 59 months with cough, difficult breathing and chest indrawing
* Written informed consent from the caretaker

Exclusion Criteria:

* Children with known heart disease
* Children on medication with Zinc supplements
* Children with obstructive air way disease
* Children with active measles
* Known intolerance or allergy to zinc or zinc-containing products

Ages: 6 Months to 59 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 328 (Estimated)
Dates: Start 2006-09; Primary Completion 2007-03 (Actual); Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
Time taken for normalisation of respiratory rate
Time taken for normalisation of Temperature
Time taken for oxygen saturation to normalise

SECONDARY OUTCOMES:
Proportion of study children who will die during the follow up period
Proportion of children who develop drug adverse effects

CONTACTS AND LOCATIONS:
Overall Officials: Maheswari s Gurusamy, MBBS, Principal Investigator — Department of Paediatrics and Child Health Makerere University, Kampala, Uganda
Locations (1):
- Department of Paediatrics and Child Health, Makerere University, Kampala, Kampala, Uganda

REFERENCES:
- [Background] Brooks WA, Yunus M, Santosham M, Wahed MA, Nahar K, Yeasmin S, Black RE. Zinc for severe pneumonia in very young children: double-blind placebo-controlled trial. Lancet. 2004 May 22;363(9422):1683-8. doi: 10.1016/S0140-6736(04)16252-1. PMID 15158629
- [Background] Bose A, Coles CL, Gunavathi, John H, Moses P, Raghupathy P, Kirubakaran C, Black RE, Brooks WA, Santosham M. Efficacy of zinc in the treatment of severe pneumonia in hospitalized children <2 y old. Am J Clin Nutr. 2006 May;83(5):1089-96; quiz 1207. doi: 10.1093/ajcn/83.5.1089. PMID 16685051
- [Background] Bitarakwate E, Mworozi E, Kekitiinwa A. Serum zinc status of children with persistent diarrhoea admitted to the diarrhoea management unit of Mulago Hospital, Uganda. Afr Health Sci. 2003 Aug;3(2):54-60. PMID 12913795
- [Background] Mahalanabis D, Lahiri M, Paul D, Gupta S, Gupta A, Wahed MA, Khaled MA. Randomized, double-blind, placebo-controlled clinical trial of the efficacy of treatment with zinc or vitamin A in infants and young children with severe acute lower respiratory infection. Am J Clin Nutr. 2004 Mar;79(3):430-6. doi: 10.1093/ajcn/79.3.430. PMID 14985218
- [Derived] Srinivasan MG, Ndeezi G, Mboijana CK, Kiguli S, Bimenya GS, Nankabirwa V, Tumwine JK. Zinc adjunct therapy reduces case fatality in severe childhood pneumonia: a randomized double blind placebo-controlled trial. BMC Med. 2012 Feb 8;10:14. doi: 10.1186/1741-7015-10-14. PMID 22316073